CLINICAL TRIAL: NCT04406883
Title: Effects of Simvastatin in the Prevention of Pain Experienced After Tooth Extraction. Double-blind Clinical Trials
Brief Title: Effects of Simvastatin in the Prevention of Pain Experienced After Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, director,clinical research, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2093
Record Dates: First submitted 2020-03-22; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Pain
Keywords: Pain Measurement;Tooth Extraction;Simvastatin.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study is a Double-blind, Randomized, Parallel-group, split-mouth.
Who Masked: Participant
Masking Description: This event was a double-blind study (neither the patients nor the clinicians were aware of the rinsing solution used). Consequently, all periods of treatment, clinical parameters were recorded by an examiner who was blinded to the kind of medication received by the subjects while another clinician gave treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A (Simavastatin 10 mg with gelatin sponge graft) (Active Comparator): A group: After atraumatic extraction, filled the tooth socket with Simvastatin10 mg solution impregnated gelatin sponge.
  Interventions: Drug: Extraction + filled with Simvastatin solution impregnated gelatin sponge
- B(Gelatin sponge graft ) (Active Comparator): B group: Following atraumatic extraction, put in the tooth socket with gelatin sponge.
  Interventions: Drug: Extraction + filled with Simvastatin solution impregnated gelatin sponge

INTERVENTIONS:
Drug: Extraction + filled with Simvastatin solution impregnated gelatin sponge — All two first premolars were extracted carefully, have used periotome as a means of atraumatic extraction that facilitated the removal of teeth with minimum damage to the surrounding alveolar bone, teeth to be extracted should have minimum periapical changes radiographically; with decreasing soft tissue reflection; the socket was tan gently irrigated with normal saline and hemostasis was achieved. It must be noted that A group (Extraction + filled with Simvastatin (Poursina Pharmaceutical Co. Tehran-Iran) solution impregnated gelatin sponge (Maquira Industry Dental Products S.A. Brazil) and B group (Extraction + without Simvastatin solution impregnated gelatin sponge), was placed in one of the sockets.
  Other Names: Extraction + filled gelatin sponge

SUMMARY:
Atraumatic extraction of maxillary premolar teeth (on the Right, left side) was done; Subsequently, the patients were randomly divided into two equal groups: A group (Extraction + filled with a Simvastatin solution impregnated gelatin sponge) and B group (Extraction + without Simvastatin solution impregnated gelatin sponge), were placed in one of the sockets; the pain level is recorded according to the VAS scores at the intervals of before treatments, also Postoperative analog pain scores were assessed in 30 minutes, 6 hours, 12 hours and 24 hours.

DETAILED DESCRIPTION:
The method of procedure was performed by the same surgeon under local anesthesia (Lidocaine 2% with epinephrine 1:100,000, made by Darou Pakhsh Pharmaceutical Co; Tehran-Iran) to avoid bias. All two first premolars were extracted carefully, have used periotome as a means of atraumatic extraction that facilitated the removal of teeth with minimum damage to the surrounding alveolar bone, teeth to be extracted should have minimum periapical changes radiographically; with decreasing soft tissue reflection; the socket was tan gently irrigated with normal saline and hemostasis was achieved. It must be noted that A group (Extraction + Simvastatin filled with Simvastatin (Poursina Pharmaceutical Co. Tehran-Iran) solution impregnated gelatin sponge (Maquira Industry Dental Products S.A. Brazil) and B group (Extraction + without Simvastatin solution impregnated gelatin sponge), was placed in one of the sockets.

ELIGIBILITY:
Inclusion Criteria:

Healthy patients Age group 18-35 years Sulcular probing not more than 3 mm and no redness The determination for extraction of teeth (two maxillary first premolars)for orthodontic treatment A tooth requiring an atraumatic extraction technique.

Exclusion Criteria:

Systemic diseases Smoking habits; pregnancy or breastfeeding Periodontitis; Teeth having radiographically obvious large periapical Lesion(abscess/granuloma/cyst) T the history of Chemotherapy Radiation therapy Periodontal and the use of any medicine (antibiotics; steroids; non-steroidal anti-inflammatory drugs Allergy to Simvastatin.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Pain experienced by patients following the atraumatic tooth extraction, evaluated by using a visual analog pain scale within 24 hours. | one day
  The pain level is recorded according to the visual analogue scale (VAS) at the intervals of before treatments, also Postoperative analog pain scores were assessed in 30 minutes to 24 hours later.

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
will published